CLINICAL TRIAL: NCT04241562
Title: Validation of a Novel Cortical Biomarker Signature for Pain
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, David Seminowicz, Associate Professor, University of Maryland, Baltimore
Other Study IDs: 1R61NS113269-01 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: TMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Injection of Nerve Growth Factor — Injection of Nerve Growth Factor to the right masseter

SUMMARY:
The study aims to undertake analytical validation of an brain biomarker in healthy participants experiencing a model of sustained temporomandibular pain. The biomarker could detect participants at greater risk of developing more severe pain.

DETAILED DESCRIPTION:
Chronic pain is a major health burden associated with immense economic and social costs. Predictive biomarkers that can identify individuals at risk of developing severe and persistent pain, which is associated with worse disability and greater reliance on opioids, would promote aggressive, early intervention that could halt the transition to chronic pain. The investigative team has uncovered evidence of a unique cortical biomarker signature that predicts pain susceptibility (severity and duration). The biomarker signature combines resting state sensorimotor peak alpha frequency (PAF) measured using electroencephalograph (EEG) and corticomotor excitability (CME) measured using transcranial magnetic stimulation (TMS). This PAF/CME biomarker signature could be capable of predicting the severity of pain experienced by an individual minutes to months in the future, as well as the duration of pain (time to recovery). In the current study, the investigators aim to undertake analytical validation of this biomarker in healthy participants using a standardized model of the transition to sustained myofascial temporomandibular pain (masseter intramuscular injection of nerve growth factor). The investigators will record PAF/CME at multiple time points before and during the development of pain and use online diaries and in-laboratory assessments of pain, sleep, stress, and other psychosocial variables. Specifically, the investigators will test if the biomarker signature predicts an individual's pain sensitivity (high- or low-pain sensitive).

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* unable or refusal to provide written consent
* presence of any acute pain disorder
* history or presence of any chronic pain disorder
* history or presence of any other medical or psychiatric compliant
* use of opioids or illicit drugs in the past 3 months
* pregnant or lactating women
* excessive alcohol use
* contraindicated for TMS (metal implants, epilepsy)

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women with no medical complaints, no history of chronic pain and no current acute pain between the ages of 18 and 44 years will be included.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Peak pain intensity from diary ratings | 0 to 30 days following NGF injection
  Pain sensitivity

SECONDARY OUTCOMES:
Average Peak daily pain intensity from from diary ratings | 0 to 30 days following NGF injection
  Pain severity
The time between pain onset and complete resolution of pain for two consecutive days | 0 to 30 days following NGF injection
  Pain duration

CONTACTS AND LOCATIONS:
Overall Officials: David A Seminowicz, PhD, Principal Investigator — University of Maryland School of Dentistry; Siobhan M Schabrun, PhD, Principal Investigator — Neuroscience Research Australia; University of New South Wales
Locations (2):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States
- Neuroscience Research Australia, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data will be made available immediately following publication via an open-access data repository.

REFERENCES:
- [Derived] Seminowicz DA, Bilska K, Chowdhury NS, Skippen P, Millard SK, Chiang AKI, Chen S, Furman AJ, Schabrun SM. A novel cortical biomarker signature for predicting pain sensitivity: protocol for the PREDICT longitudinal analytical validation study. Pain Rep. 2020 Jul 27;5(4):e833. doi: 10.1097/PR9.0000000000000833. eCollection 2020 Jul-Aug. PMID 32766469